CLINICAL TRIAL: NCT00337051
Title: Sevoflurane-induced Prevention of Ischemia-reperfusion Lesions in Renal Allograft Transplants Recipients
Brief Title: Renal Transplantation and Inhaled Anesthetic Sevoflurane (SEVOREIN)
Acronym: SévoRein
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9413-04; 2003-048
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: End-stage Chronic Renal Disease; Severe Acute Kidney Failure; Renal Transplantation
Keywords: Renal transplantation; renal allograft; end-stage renal disease; renal failure; general anaesthesia; inhaled anaesthetic; Sevoflurane; ischemia; reperfusion; ischemic lesions
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Renal Insufficiency; Ischemia | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S (Experimental): General Anesthesia with sevoflurane (inhalation) as hypnotic
  Interventions: Drug: Sevoflurane
- P (Active Comparator): General Anesthesia With Propofol TCI
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — General anesthesia using Sevoflurane (inhalation) as hypnotic
  Arms: S
Drug: Propofol — General anesthesia with propofol TCI
  Arms: P

SUMMARY:
Renal transplantation is characterized by ischemia-reperfusion lesions in allograft. In a previous study, Julier and al. (Anesthesiology 2003) have demonstrated that sevoflurane reduces glomerular lesions in kidney of patients undergoing a cardiovascular surgery and présenting with ischemia-reperfusion phenomena.

The purpose of the study is to evaluate the effects of sevoflurane on the recovery of renal graft function in patients after kidney transplantation.

This study will be a randomized, double blinded, controlled clinical trial and 120 patients undergoing renal allograft transplantation will be included.

Patients will be divided into 2 groups: one group of patients who will receive sevoflurane (evaluated treatment) for anaesthesia and the other one who will receive propofol (reference treatment).

We will evaluate renal function for one year after transplantation. Ours results will confirm or not that sevoflurane protects kidney function from ischemia-reperfusion lesions.

DETAILED DESCRIPTION:
Introduction :

Renal transplantation is characterized by ischemia-reperfusion lesions in allografts. Prolonged cold ischemia duration, age of donor (older than 50) or donor cardiac arrest are common factors associated with delayed graft function. In cardiac surgery, Sevoflurane (a volatile-inhaled anesthetic) protects the heart from ischemia-reperfusion lesions and preserves glomerular filtration function in patients. This cardioprotective effect involves K+-ATP mitochondrial channels which are also known to be expressed in renal cells.

Therefore, it is interesting to evaluate Sevoflurane effects in the context of renal allograft transplantation in order to shorten the delayed graft function and enhance post-operative renal function

Objectives:

Main goal:

Evaluate time necessary to obtain serum creatinine levels inferior to 200µmol/l of the recipient in the group receiving Sevoflurane in comparison with the group of patients receiving propofol infusion for general anaesthesia

Secondary goals:

* Compare serum creatinine levels in the two groups at day14
* Compare patient survival and acute rejection occurrence over a period of one-year follow-up in the two groups
* Compare the safety of both anesthetics assessed as renal tubular injury-toxicity (by measuring serum levels of NAG) and levels of serum inorganic fluor products in the post-operative period; and by referencing all adverse events
* Compare the effect of both anesthetics on delayed-recovery graft function by assessing clinical end-points (daily diuresis, number of haemodialysis sessions in the two weeks following transplantation) and biological end-points (serum creatinin and cystatinC levels in the two weeks following transplantation)

Patients:

120 patients scheduled to undergo a renal allograft transplantation with transplants defined by either a cold ischemia duration of more than 20h or a donor's age older than 50 years or a donor cardiac arrest will be randomized in 2 groups of sixty patients undergoing two different general anesthesia protocols. All patients will be included in the Renal Transplantation Unit of Bordeaux University Hospital, Aquitaine, France.

Methods:

This study will be a clinical randomized trial on 2 parallel groups. It will be double-blind for nephrologists and biologists who evaluate the end-points and will involve a population of renal transplanted patients.

The study will compare clinical and biological outcomes according to the type of general anesthesia undergone for transplantation:

* One group of patients with inhaled anesthesia by Sevoflurane (evaluated treatment)
* One group of patients with intravenous anesthesia by propofol (reference treatment).

Patients will be evaluated over a period of one year follow-up. This study is multicentric, based in Aquitaine for a period of three years, involving anaesthesiologists, nephrologists, and urologists.

Baseline brain-dead donor and graft donation characteristics will be collected by the Hospital Coordination team in Bordeaux, Pau and Bayonne.

Statistical analysis will be on intention-to-treat basis. Expected results: 1-Demonstrate Sevoflurane benefit for ischemia-reperfusion protection in renal allograft and a shortened recovery of renal graft function in the two-week post-operative period in the group allocated for Sevoflurane exposure during anaesthesia. 2-Confirm the good safety of Sevoflurane exposure in chronic end-stage renal diseased patients undergoing renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* scheduled to undergo renal allograft transplantation
* transplant : cold ischemia duration > 20 hours or donor age > 50 years or donor cardiac arrest
* ASA 2-3
* social security affiliation
* informed consent signed

Exclusion Criteria:

* halogenated anesthetic agent hypersensibility
* medical history or familial history of malignant hyperthermia
* porphyria
* pregnancy or breast feeding
* hyperimmunized patient
* participation in an immunosuppressive drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-06; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
time to obtain serum creatinine levels inferior to 200µmol/l in the transplant recipient | evalued at 14 days

SECONDARY OUTCOMES:
creatinemia levels at day 14 | evalued at 14 days
patient survival | during 1 year follow-up
acute rejection occurrence | during 1 year follow-up
safety : renal tubular injury toxicity (serum cystatinC and NAG), serum inorganic fluor products | 1, 2 and 3 days after kidney transplantation
other clinical end-points: daily diuresis, number of haemodialysis sessions | during the two weeks following transplantation
other biological end-points: serum creatinin and cystatinC levels | during the two weeks following transplantation
Other adverse events | during one year folow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francois SZTARK, Pr, Principal Investigator — University Hospital, Bordeaux; Paul PEREZ, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Département d'anesthésie réanimation 1 - Hôpital Pellegrin - CHU de Bordeaux, Bordeaux, France